CLINICAL TRIAL: NCT00368199
Title: Diagnostic Value Transcranial Duplex Scanning and Single Photon Emission Tomography in Patients Suspected of Having Idiopathic Parkinson Disease or Atypical Parkinson Syndromes
Brief Title: Transcranial Duplex Scanning and Single Photon Emission Computer Tomography (SPECT) in Parkinsonian Syndromes
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Funding: Stichting Internationaal Parkinson Fonds, The Netherlands (Unknown)
Responsible Party: Principal Investigator, Wim Weber, Associate Professor of Neurology, Maastricht University Medical Center
Other Study IDs: 1-Vlaar
Record Dates: First submitted 2006-08-22; First posted 2006-08-24 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Parkinson's Disease; Parkinsonian Syndrome; Multiple System Atrophy; Supranuclear Palsy, Progressive; Essential Tremor; Vascular Parkinsonism; Drug Induced Parkinsonism
Keywords: single photon emission computer tomography (SPECT); transcranial sonography; transcranial duplex scanning; parkinson's disease; atypical parkinson syndromes; parkinsonism; parkinsonian; diagnostic; progressive supranuclear paralysis
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Multiple System Atrophy; Supranuclear Palsy, Progressive; Essential Tremor; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — no biocpsicmens
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study is to determine the sensitivity and specificity of transcranial duplex scanning (TCD) and single photon emission computer tomography (SPECT) in patients suspected of having Idiopathic Parkinson Disease (PD) or Atypical Parkinson Syndromes (APS) with as golden standard the clinical diagnosis after 2-year follow-up.

DETAILED DESCRIPTION:
PD is a progressive neurodegenerative illness that affects about 50.000 people in the Netherlands. Diagnosis is based on clinical criteria. However, purely on clinical grounds, especially in the early stage, it is not possible to differentiate PD from other parkinsonian syndromes like multiple system atrophy, Progressive Supranuclear Palsy, vascular parkinsonism, drug induced parkinsonism and essential tremor. Accurate differentiation is important because treatment and prognosis varies between the different syndromes.

At present SPECT scans are used mostly. However the SPECT is only used in the minority of the patients suspected of PD mainly because the costs and the discussion about their sensitivity and specificity to diagnose PD. We are currently finishing a meta-analysis on the diagnostic value of the SPECT in patients with parkinsonian diseases.

Recently an alternative method to visualise the alterations in the cerebral dopaminergic pathways of PD patients has been proposed: TCD of the substantia nigra in the brainstem. This technique has high inter-observer reliability. Becker discovered in 1994 that patients with PD had bilateral hyperechogenicity of the substantia nigra. Neuropathological studies confirm the increased echogenicity is because of iron deposition. However the reason of the increased level of iron is unknown.

Several publications confirm the observation that up to 90% of PD patients have increased echogenicity of the substantia nigra. In healthy subjects and in patients with essential tremor this hyperintensity of the substantia nigra is only found in 10%. However 60% of the healthy subjects with increased echogenicity also have decreased nigra-striatal function on (18)-F-dopa-PET. So TCD might possibly be an early (presymptomatic) marker for PD.

If substantia nigra scanning is combined with scanning of the nucleus lentiformis, the differentiation between PD and APS is increased. Another advantage is that with the same technique the raphe nuclei can be made visible. Several studies confirm the echogenicity of raphe nuclei is decreased in PD patients with a depression.

Our own experience suggests that the positive predictive value of this technique nears that of SPECT scans. In our pilot study with 45 patients with PD or APS who underwent SPECT and TCS we found a positive prediction value of 95%. This would predict that, if TCE is compatible with PD, a SPECT does not provide additional information; so in theory one might reduce the amount of SPECT's in almost 50% of cases.

A direct compare of the diagnostic accuracy as to PD between duplex and SPECT scans has until now not been made. Our hypothesis is that the TCD of substantia nigra duplex scanning is an accurate diagnostic tool and deserves a place in the diagnostic work-up of PD/Parkinsonism patients and diagnostically efficient enough to replace 50% of SPECT scans. In comparison with SPECT duplex scanning is less costly (respectively 80 euro and 400 euro for each SPECT) and more comfortable for the patient.

Methods:

Subjects:

250 consecutive patients with new parkinsonian complaints in the out-patient clinic of our university hospital (Maastricht) and a local hospital.

Study design:

The investigator will give a clinical diagnosis at the first visit. All subjects undergo SPECT and duplex scanning, both tests will be judged blindly for the clinical diagnosis. After two years follow-up, all patients will be seen by the investigator and again a clinical diagnosis will be made (investigator is blinded for the results of the duplex and SPECT). At the end of the follow-up the sensitivity and specificity of the first clinical judgement, duplex and SPECT can be calculated. The golden standard is the clinical diagnosis at the end of the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unclear parkinsonism at the outpatient clinic

Exclusion Criteria:

* Known diagnosis at presentation
* Life expectation of less than two years because of a non neurological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 250 Patients with unclear parkinsonism at the outpatient clinic
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2006-09-01 (Actual); Primary Completion 2008-09-18 (Actual); Study Completion 2012-09-15 (Actual)

PRIMARY OUTCOMES:
Concordance of hyperechogenic SN with clinical diagnosis of Parkinson's | 24 months
  Hyperechogenic substabtia nigra (SN) was assessed at initial visit and after 2 years, patients were re-examined by two movement disorder specialist neurologists for a final clinical diagnosis that served as a surrogate gold standard for our study.

CONTACTS AND LOCATIONS:
Overall Officials: Wim EJ Weber, MD PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, PO Box 5800, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Dataset is published with PeerJ
Time Frame: Is availabel
Access Criteria: Publicly available
URL: https://peerj.com/articles/2037

REFERENCES:
- [Result] Bouwmans AE, Vlaar AM, Mess WH, Kessels A, Weber WE. Specificity and sensitivity of transcranial sonography of the substantia nigra in the diagnosis of Parkinson's disease: prospective cohort study in 196 patients. BMJ Open. 2013 Apr 2;3(4):e002613. doi: 10.1136/bmjopen-2013-002613. Print 2013. PMID 23550093
- [Result] Bouwmans AE, Leentjens AF, Mess WH, Weber WE. Abnormal Echogenicity of the Substantia Nigra, Raphe Nuclei, and Third-Ventricle Width as Markers of Cognitive Impairment in Parkinsonian Disorders: A Cross-Sectional Study. Parkinsons Dis. 2016;2016:4058580. doi: 10.1155/2016/4058580. Epub 2016 Jan 10. PMID 26881179
- [Result] Bouwmans AE, Weber WE, Leentjens AF, Mess WH. Transcranial sonography findings related to depression in parkinsonian disorders: cross-sectional study in 126 patients. PeerJ. 2016 May 18;4:e2037. doi: 10.7717/peerj.2037. eCollection 2016. PMID 27231659
- [Derived] Vlaar AM, Bouwmans AE, van Kroonenburgh MJ, Mess WH, Tromp SC, Wuisman PG, Kessels AG, Winogrodzka A, Weber WE. Protocol of a prospective study on the diagnostic value of transcranial duplex scanning of the substantia nigra in patients with parkinsonian symptoms. BMC Neurol. 2007 Sep 4;7:28. doi: 10.1186/1471-2377-7-28. PMID 17784944
- See also: Sponsorship — http://parkinsonfonds.nl
- Available data/document: Individual Participant Data Set — https://peerj.com/articles/2037/